CLINICAL TRIAL: NCT06169189
Title: The Effect of Education Given to Nursing Students on Their Environmental Attitudes: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Hasan EVCİMEN, RN, PhD, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 05.10.23/8-19
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Nursing Student

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention group (Active Comparator): The experimental group will be given 8-week global warming-climate change based training
  Interventions: Behavioral: global warming-climate change based education
- Control Group (No Intervention): The initiative will not be implemented.

INTERVENTIONS:
Behavioral: global warming-climate change based education — The experimental group will be given 8 weeks of global warming-climate change based training. No intervention will be applied to the control group.
  Arms: Experimental intervention group

SUMMARY:
This study is conducted to examine the effect of climate change and global warming-based education given to nursing students on their environmental attitudes. The research was planned as a randomized controlled experimental. According to the posthoc power analysis, it was determined that the type one error amount was 0.05 with a medium effect size and the power of the study was 94% when 110 participants were taken. The data were included from the 2nd, 3rd and 4th grades of a nursing faculty in eastern Turkey. Assignments were made to experimental and control groups by randomization. Personal information form and environmental attitude scale were used to collect data.

DETAILED DESCRIPTION:
Climate change and global warming are a global public health problem. This situation, which affects all masses, also deeply affects human life. Future nurses need to have high awareness of this situation and educate and inform the society about this situation. Nurse students' environmental attitudes, knowledge and behavior towards the environment need to be increased. The aim of this research is to determine the effect of global warming and climate change-based education given to nursing students on their environmental attitudes.The research was planned as a randomized controlled experimental. According to the posthoc power analysis, it was determined that the type one error amount was 0.05 with a medium effect size and the power of the study was 94% when 110 participants were taken. The data were included from the 2nd, 3rd and 4th grades of a nursing faculty in eastern Turkey. Assignments were made to experimental and control groups by randomization. Personal information form and environmental attitude scale were used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in research
* have verbal communication skills

Exclusion Criteria:

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
change of environmental attitude scale | baseline to 2 months
  environmental attitude scale; It was developed by Berberoğlu and Tosunoğlu to determine the environmental attitudes of university students. The scale is a 5-point Likert type and consists of 21 items. The scale contains 11 reverse items. These items are reverse coded. It is stated that the Cronbach alpha of the scale is 0.77.

CONTACTS AND LOCATIONS:
Locations (1):
- Muş Alparslan University, Muş, Turkey (Türkiye)

REFERENCES:
- [Derived] Evcimen H, Ciftci N, Yildiz M. Effect of Environmental Awareness-Based Education on Environmental Attitudes of Nursing Students: A Randomized Controlled Study. Public Health Nurs. 2025 Jan-Feb;42(1):411-418. doi: 10.1111/phn.13426. Epub 2024 Oct 7. PMID 39375322